CLINICAL TRIAL: NCT00399893
Title: Investigation of the Developmental, Nutritional and Hormonal Regulation of Ghrelin in Children and Young Adults With Prader-Willi Syndrome (PWS): Octreotide Intervention Sub-study
Brief Title: Octreotide Therapy in Children and Young Adults With Prader-Willi Syndrome (PWS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00005426; Protocol #00005426 (Other Grant/Funding Number: NIH:1K23-RR021979, GCRC M01-RR-30 (NCRR))
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-06

CONDITIONS: Prader-Willi Syndrome
Keywords: Childhood obesity; Prader-Willi Syndrome; Octreotide; Ghrelin; Weight loss; Body composition; Energy expenditure
MeSH Terms: conditions — Prader-Willi Syndrome; Pediatric Obesity; Weight Loss | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Octreotide (Experimental): Octreotide to be administered by subcutaneous injection three times daily while on study
  Interventions: Drug: Octreotide
- Placebo (Placebo Comparator): Placebo to be administered by subcutaneous injection three times daily while on study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Octreotide — Octreotide to be administered by subcutaneous injection three times daily
  Other Names: Sandostatin
  Arms: Octreotide
Drug: Placebo — Placebo to be administered by subcutaneous injection three times daily while on study
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate over a 6 month period the effect of octreotide therapy on food intake, sense of hunger, body weight, body composition, efficiency of burning calories, biomarkers of weight regulation and growth hormone markers in children and young Adults with Prader-Willi Syndrome(PWS).

DETAILED DESCRIPTION:
Obesity continues to be a prevalent health concern affecting every race of the American population. According to data from the World Health Organization, 54% of U.S. adults are overweight (body mass index (BMI) >25 kg/m2 ) and 22% are obese (BMI >30 kg/m2) (1). In addition, 25% of U.S. children are overweight or obese (1). Studies show that obese children are likely to become obese adults (2-5). Also, recent studies report significant years of life lost due to the impact of being an obese adult (6, 7). Thus, insights into the pathogenesis of childhood obesity and preventative measures are needed to combat the inevitable increase in worldwide incidence of obesity and its associated co-morbidities. Recent studies have identified a new gastroenteric hormone, ghrelin, as a long-term regulator of energy balance in humans (12). Ghrelin is a 28 amino acid acylated peptide which is an endogenous ligand of the growth hormone secretagogue receptor (GHS-R), a hypothalamic G-protein-coupled receptor (13). Enteroendocrine cells (X/A-like cells) of the stomach are the major site of ghrelin synthesis, although a minor proportion of ghrelin synthesis occurs in other sites such as the hypothalamus, pituitary, duodenum, jejunum and lung (14) (15, 16).

The hypothesis that hyperghrelinemia causes some of the features of PWS predicts that this disorder will be ameliorated (partially or completely) by lowering ghrelin levels. We have recently shown that the somatostatin agonist, octreotide, suppresses ghrelin levels in humans. If octreotide remains effective in longer term studies, the drug may become an adjuvant therapy, in addition to growth hormone, to control the insatiable appetite and morbid obesity seen in this condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PWS confirmed by chromosome analysis
* Ages 5 years to 21 years
* BMI for age ≥ (greater-than or equal to)85th percentile
* Written informed consent and assent obtained and willingness to comply with the study schedule and procedures
* Free T4, Thyroid stimulating hormone (TSH) values in the normal range (either endogenous or with thyroxine replacement)

Exclusion Criteria:

* Patients with any other clinically significant disease that would have an impact on body composition, including diabetes mellitus, chronic inflammatory bowel disease, chronic severe liver or kidney disease or neurologic disorders
* Concomitant use of an investigational drug or Octreotide in the past year
* Use of steroids for longer than 7 days within the past 30 days

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Haqq, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Haqq AM, Stadler DD, Rosenfeld RG, Pratt KL, Weigle DS, Frayo RS, LaFranchi SH, Cummings DE, Purnell JQ. Circulating ghrelin levels are suppressed by meals and octreotide therapy in children with Prader-Willi syndrome. J Clin Endocrinol Metab. 2003 Aug;88(8):3573-6. doi: 10.1210/jc.2003-030205. PMID 12915638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for the study were recruited over a period of 2.5 years. Participants were identified from the medical clinics or from IRB approved advertisements.
Pre-assignment Details: Participants were eligible to enroll into the study with a diagnosis of PWS proven by chromosome analysis and thyroid function tests within normal ranges. Participants could not have used the study drug within the past year and could not have been on steroids within the past 30 days. These items would exclude participation.
Groups:
- Octreotide: Octreotide :
  Octreotide : Octreotide or placebo to be administered by subcutaneous injection three times daily
- Placebo Comparator: Placebo to be administered by subcutaneous injection three times daily while on study
Period: Overall Study
Arm/Group | Octreotide | Placebo Comparator
Started | 2 | 3
Completed | 1 (Participant withdrew after 3 months but was included in results) | 3
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide | Placebo Comparator | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 5
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11 (4.2) | 13 (4.6) | 11.8 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Decrease in Fasting Total Ghrelin
Description: Number of participants showing a decrease in Fasting total ghrelin from baseline to 6 months of treatment with Octreotide or placebo
Time Frame: 6 months
Population: Descriptive statistics or percent of change from the baseline for the 5 patients was used.
  A patient withdrew but included in analysis.
Measure: Number; unit: Participants
Arm/Group | Octreotide | Placebo Comparator
Number analyzed (Participants) | 2 | 3
Participants | 1 | 1

2. Secondary Outcome: Number of Participants With Decreased Body Composition From Baseline to 6 Months by BOD POD®
Description: Number of participants with decreased body-composition as Measured by BOD POD® body composition tracking system from baseline to 6 months of Octreotide or Placebo therapy
Time Frame: 6 months
Population: Participant withdrew but data was used for analysis
Measure: Number; unit: participants
Arm/Group | Octreotide | Placebo Comparator
Number analyzed (Participants) | 2 | 3
participants | 2 | 3

3. Primary Outcome: Number of Participants With Decrease in Weight From Baseline to 6 Months
Description: Number of participants who had a decrease in weight from baseline to 6 months of Octreotide or placebo therapy
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Octreotide | Placebo Comparator
Number analyzed (Participants) | 2 | 3
participants | 0 | 2

4. Primary Outcome: Number of Participants With Decreased BMI Z-score From Baseline to 6 Months
Description: Number of participants with decreased BMI z-score from baseline to 6 months of Octreotide or Placebo therapy
Time Frame: 6 months
Population: A participant withdrew but was included in analysis
Measure: Number; unit: participants
Arm/Group | Octreotide | Placebo Comparator
Number analyzed (Participants) | 2 | 3
participants | 0 | 2

5. Primary Outcome: Number of Participants With Decreased Skin-fold Measurements From Baseline to 6 Months
Description: Number of participants with decreased skin-fold measurements from baseline to 6 months of Octreotide or Placebo therapy
Time Frame: 6 months
Population: The skin fold measurements were performed; however, the data was not completed in a manner that could be analyzed; therefore we could not analyze the data. Completed data is not available to complete this outcome.
Arm/Group | Octreotide | Placebo Comparator
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Number of Participants With Decrease in Hunger and Food Intake
Description: Measured by hunger and hyperphagia by questionnaires and parent-reported 72-hour food recall from baseline to 6 months. Multiple questionnaires consisting of a battery of free text answer questions and food diaries are combined in order to make a behavioral assessment of the participants food state of hunger and food intake. There is no defined scale for this assessment. Each participants responses and parent responses are combined.
Time Frame: 6 months
Population: For this outcome measure, data from questionnaires and forms was not completed. Data for all questionnaires is not available to report.
Arm/Group | Octreotide | Placebo Comparator
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Decreased Body-composition From Baseline to 6 Months by DEXA
Description: Number of participants with decreased body-composition as Measured by Dual Energy X-ray Absorptiometry (DEXA) scan from baseline to 6 months of Octreotide or Placebo therapy
Time Frame: 6 months
Population: Data for this outcome was not analyzed
Measure: Number; unit: participants
Arm/Group | Octreotide | Placebo Comparator
Number analyzed (Participants) | 2 | 3
participants | 0 | 0

8. Primary Outcome: Number of Participants With Improved Insulin Regulation From Baseline to 6 Months
Description: Number of participants with improved Insulin regulation from baseline to 6 months of Octreotide or Placebo therapy. Insulin regulation was measured by immunochemiluminescent assay.
Time Frame: 6 months
Population: Participant withdrew but was used in the data analysis
Measure: Number; unit: participants
Arm/Group | Octreotide | Placebo Comparator
Number analyzed (Participants) | 2 | 3
participants | 2 | 0

9. Primary Outcome: Number of Participants With Improved Adiponectin Regulation From Baseline to 6 Months
Description: Number of participants with improved Adiponectin regulation from baseline to 6 months of Octreotide or Placebo therapy
Time Frame: 6 months
Population: A participant withdrew but data was used for analysis
Measure: Number; unit: participants
Arm/Group | Octreotide | Placebo Comparator
Number analyzed (Participants) | 2 | 3
participants | 2 | 2

10. Primary Outcome: Number of Participants With Improved Leptin Regulation From Baseline to 6 Months
Description: Number of participants with improved Leptin regulation from baseline to 6 months of Octreotide or Placebo therapy
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Octreotide | Placebo Comparator
Number analyzed (Participants) | 2 | 3
participants | 1 | 2

11. Primary Outcome: Number of Participants With Improved Peptide YY (PYY) Regulation From Baseline to 6 Months
Description: Number of participants with improved Peptide YY (PYY) regulation from baseline to 6 months of Octreotide or Placebo therapy
Time Frame: 6 months
Population: Participant withdrew but data was used for analysis
Measure: Number; unit: participants
Arm/Group | Octreotide | Placebo Comparator
Number analyzed (Participants) | 2 | 3
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event collection began with administration of study drug or placebo and concluded 30 days after discontinuation of study drug.
Arm/Group | Octreotide | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octreotide (N=2) | Placebo Comparator (N=3)
Gallstones (Gastrointestinal disorders) | 0 (0) | 1 (1) — One patient in the placebo group developed a small gallstone at 6 months; all patients in the active treatment group maintained normal gallbladder ultrasounds at 6 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less